CLINICAL TRIAL: NCT05471947
Title: Use of TCA 15% + 3% Glycolic Acid Chemical Peel for Improvement in Hand Lentigines
Brief Title: TCA 15% Chemical Peel for Improvement in Hand Lentigines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Main Line Center for Laser Surgery (Other)
Responsible Party: Principal Investigator, Kachiu Lee, MD, Principal Investigator, Main Line Center for Laser Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC20220721
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Photoaging; Lentigo
Keywords: Photoaging; Chemical Peel; Lentigines; Hand Rejuvenation
MeSH Terms: conditions — Lentigo | interventions — Trichloroacetic Acid; glycolic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Treatment of hand lentigines with 15% trichloroacetic acid + 3% glycolic acid
  Interventions: Drug: 15% Trichloroacetic acid + 3% glycolic acid

INTERVENTIONS:
Drug: 15% Trichloroacetic acid + 3% glycolic acid — Treatment of the hand with an over-the-counter chemical peel containing 15% trichloroacetic acid + 3% glycolic acid
  Other Names: 15% TCA + 3% GA

SUMMARY:
This study will evaluate the efficacy of the a 15% trichloroacetic acid + 3% glycolic acid peel combination for treatment of lentigines on the hands. This peel combination is sold over the counter. Patients will receive 3 treatments (spaced 4 weeks).

DETAILED DESCRIPTION:
This clinical investigation is a prospective study consisting of a screening visit, 3 treatment visits, and 1 follow-up visit. Baseline and post-treatment photos will be graded and compared.

A total of 20 patients will be recruited. Following informed consent and screening, subjects' dorsal hands will be photographed.

Patients will receive 3 treatments with the 15% TCA + 3% glycolic acid peel every 4-6 weeks on the dorsal hands. Post-treatment, patients will be instructed to apply Aquaphor to the treated area twice daily for 5 days. Patients' hands will be photographed at each visit.

Four to six weeks after their final treatment, subjects will return for photography.

ELIGIBILITY:
Inclusion Criteria:

* Age >21
* No laser, chemical peel, neuromodulator, filler treatment to the hands in >3 months
* At least 5 lentigines on each hand

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Allergy to trichloroacetic acid
* Allergy to glycolic acid
* Open wounds on treatment area (hands)
* Active inflammatory disease on treatment area such as atopic dermatitis, psoriasis, dermatomyositis

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Improvement in hand lentigines on a 5-point scale | 4-6 weeks after last treatment
  Photos will be graded on a 5 point scale (0=no change, 1=1-25% change, 2=26-50% change, 3=51-75% change, 4=76-100% change)

SECONDARY OUTCOMES:
Improvement in hand lentigines using the Global Aesthetic Improvement Scale | 4-6 weeks after last treatment
  The GAIS is a validated scale assessing overall change after aesthetic procedures

CONTACTS AND LOCATIONS:
Overall Officials: Kachiu Lee, MD, Principal Investigator — Main Line Center for Laser Surgery
Locations (1):
- Main Line Center for Laser Surgery, Ardmore, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cook KK, Cook WR Jr. Chemical peel of nonfacial skin using glycolic acid gel augmented with TCA and neutralized based on visual staging. Dermatol Surg. 2000 Nov;26(11):994-9. doi: 10.1046/j.1524-4725.2000.026011994.x. PMID 11096382
- [Result] Abd Elazim NE, Makboul R, Botros SN, Awad SM. Cryopeeling versus trichloroacetic acid peeling in the treatment of solar lentigines: Effect on epidermal Langerhans cells. Dermatol Ther. 2020 May;33(3):e13288. doi: 10.1111/dth.13288. Epub 2020 Mar 9. PMID 32118343
- [Result] Raziee M, Balighi K, Shabanzadeh-Dehkordi H, Robati RM. Efficacy and safety of cryotherapy vs. trichloroacetic acid in the treatment of solar lentigo. J Eur Acad Dermatol Venereol. 2008 Mar;22(3):316-9. doi: 10.1111/j.1468-3083.2007.02409.x. Epub 2007 Oct 18. PMID 18021205
- [Derived] Alajmi A, Niaz G, Chen C, Lee K. A 15% Trichloroacetic Acid + 3% Glycolic Acid Chemical Peel Series Improves Appearance of Hand Lentigines: An Evaluator-Blinded, Split-Hand Prospective Trial. Dermatol Surg. 2024 May 1;50(5):467-470. doi: 10.1097/DSS.0000000000004114. Epub 2024 Mar 8. PMID 38460193